CLINICAL TRIAL: NCT00080275
Title: An Open-Label Evaluation of the Safety and Efficacy of a Combination of Niacin ER and Simvastatin in Patients With Dyslipidemia (OCEANS)
Brief Title: Evaluation of the Safety & Efficacy of a Combination of Niacin ER & Simvastatin in Patients With Dyslipidemia (OCEANS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kos Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 019-02-03-CR; OCEANS
Record Dates: First submitted 2004-03-25; First posted 2004-03-29 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-10

CONDITIONS: Hypercholesterolemia
Keywords: Niacin; Statin; Zocor; Simvastatin; Coronary Heart Disease; Dyslipidemia; Atherosclerosis; Hypercholesterolemia; Stroke; High-Density Lipoprotein Cholesterol; Low-Density Lipoprotein Cholesterol; Lipoprotein; Lipid; Niacin ER/simvastatin; Total Cholesterol; Triglycerides
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease; Dyslipidemias; Atherosclerosis; Stroke | interventions — Simvastatin

INTERVENTIONS:
Drug: Niacin Extended-Release and simvastatin Tablets

SUMMARY:
The purpose of this 24 week study is to compare the effectiveness and safety of different doses of Niacin ER/Simvastatin (NS) in subjects with elevated fat levels in their blood (dyslipidemia).

At least 600 subjects with a similar medical condition will take part in this study.

DETAILED DESCRIPTION:
Objectives:

To evaluate the safety and efficacy of the combination product niacin ER and simvastatin (NS) in patients with primary type II dyslipidemia and to descriptively compare flushing rates between two Titration Schedules for NS.

ELIGIBILITY:
Inclusion Criteria:

* Patient has primary Type II hyperlipidemia or mixed dyslipidemia.
* If the patient is currently taking a lipid modifying medication other than Zocor & he/she is willing to discontinue this medication
* LDL-C levels and/or non HDL-C levels above normal.
* Reasonable compliance with a standard cholesterol-lowering diet for a minimum of 4 weeks prior to screening and for the duration of the study.

Exclusion Criteria:

* Patient has an allergy, hypersensitivity, or intolerance to niacin, statins, or their derivatives.
* HbA1c ≥ 9% in diabetic patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-03

REFERENCES:
- [Derived] Karas RH, Kashyap ML, Knopp RH, Keller LH, Bajorunas DR, Davidson MH. Long-term safety and efficacy of a combination of niacin extended release and simvastatin in patients with dyslipidemia: the OCEANS study. Am J Cardiovasc Drugs. 2008;8(2):69-81. doi: 10.2165/00129784-200808020-00001. PMID 18422390